CLINICAL TRIAL: NCT06868108
Title: Clinical Trial on the Effect of the Flexible Suturing System With Anchors (FSSA) in Full-thickness Rotator Cuff Tendon Tears
Status: Enrolling by invitation | Type: Observational
Sponsor: Integrity Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DN-00808
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Flexible Suturing System with Anchors (FSSA) — Surgically repaired full-thickness rotator cuff tendon tears with the Flexible Suturing System with Anchors (FSSA).

SUMMARY:
The purpose of this research study is to evaluate tendon healing when using the Flexible Suturing System with Anchors (FSSA) to surgically repair full-thickness rotator cuff tendon tears.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST meet ALL the following criteria to be included in the study:

1. Underwent surgery to repair a torn rotator cuff tear with the Flexible Suturing System with Anchors (FSSA) and is able to obtain a follow-up MRI within 12 months +4 months / -1 month from the surgery date.
2. Tear size of the supraspinatus (SSP) with or without involvement of the infraspinatus (ISP), confirmed intra-operatively or with the pre-procedural MRI, is greater than or equal to 1 cm.
3. Between 18 and 70 years old at the time of surgery.
4. Able to understand the content of the subject information / Informed Consent Form (ICF) and is willing and able to participate in the prospective data collection protocol and comply with the required data collection.

Exclusion Criteria:

Subjects will be excluded from the study if they meet ANY of the following criteria:

1. Had a prior rotator cuff surgery on the index shoulder.
2. Has a subscapularis tear with a Lafosse score of 3 or greater, or a teres minor tear requiring repair.
3. Identified as being repaired in a hybrid approach, where a non-FSSA anchor is used in the case for SSP and/or ISP rotator cuff repair.
4. SSP and / or ISP tendon ruptures that are considered irreparable or only partially repairable at the time of the intervention.
5. At any time during the previous 18 months was involved in a workers compensation case or litigation related to bodily injury, whether related or unrelated to the index shoulder.
6. Has a history of chronic opioid use.
7. Subjects with condition(s) that contraindicate or complicate outcomes of ARCR such as:

   * Current or prior infection of the ipsilateral shoulder
   * Known inflammatory arthropathy or history of inflammatory arthropathy
   * Chronic joint disease
   * Concomitant labral fixation
   * Concomitant os acromial fixation
   * Glenohumeral joint instability (multiple dislocations/subluxations)
   * Subacromial or intra-articular injection within 3 months prior to surgery
   * Oral or injected steroid use in the following timeframe: 4 weeks prior to surgery through current date
   * Hamada 3 or greater rotator cuff arthropathy on X-ray
   * Goutallier atrophy > Grade 3
   * Proximal humeral fracture or scapular fracture
   * Avascular necrosis of humeral head or glenoid
   * Immunodeficiency disorders
   * Chronic inflammatory disorders
   * Osteoarthritis >2 (Samilson-Prieto)
8. Has other concurrent medical or other conditions (chronic or acute in nature) that in the opinion of the participating investigator may prevent participation or otherwise render subject ineligible for the study.
9. Subjects who are unable to tolerate magnetic resonance imaging (MRI), due to psychiatric or medical contraindications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An individual that underwent surgery to repair a torn rotator cuff tear with the Flexible Suturing System with Anchors (FSSA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | One year
  The cumulative healing rate of the repaired rotator cuff tendon, confirmed through MRI, studied one year after the intervention and using the Sugaya classification (Sugaya H (2005)), where healing is defined as Sugaya Type I, II, or III.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Texas Orthopedic Specialist, Bedford, Texas
  - Houston Methodist The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No